CLINICAL TRIAL: NCT03014505
Title: Fecal Microbiota Transplantation Versus Standard Therapy in Decompensated Cirrhosis: A Randomized Controlled Trial
Brief Title: Fecal Microbiota Transplantation for Decompensated Cirrhosis
Acronym: FMTDC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chengdu Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMT-GYH
Record Dates: First submitted 2017-01-03; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Decompensated Cirrhosis; Fecal Microbiota Transplantation
Keywords: Cirrhosis; Fecal Microbiota Transplantation; Intestinal flora; Intestinal mucosal barrier; Intestinal Bacteria Flora Disturbance
MeSH Terms: conditions — Fibrosis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FMT (Experimental): Fecal Microbiota Transplantation via endoscope and/or cenema and the traditional treatments
  Interventions: Biological: FMT
- The traditional treatments (Active Comparator)
  Interventions: Other: traditional treatments

INTERVENTIONS:
Biological: FMT — Fecal Microbiota Transplantation and the traditional treatments for Decompensated Cirrhosis in part 1
  Other Names: Fecal Microbiota Transplantation
  Arms: FMT
Other: traditional treatments — traditional treatments for Decompensated Cirrhosis in part 2
  Arms: The traditional treatments

SUMMARY:
Imbalance of gut bacteria is suspected to play a key role driving the progression of cirrhosis and there is hope manipulation of these bacteria may be beneficial. This study will determine if fecal microbiota transplantation is an effective and safe treatment for decompensated cirrhosis.

DETAILED DESCRIPTION:
Two groups of inpatients with decompensated cirrhosis will be randomized using random sequence generator into experimental and control groups. Two groups will given traditional treatments and experimental group will added treatment with fecal microbiota transplantation via endoscope and/or cenema.The liver function parameters, adverse events complication, systemic inflammatory markers, Intestinal mucosa structure, permeability changes in the intestinal mucosal barrier, Microbiota composition will be assessed and thereafter at 1 month and 3 months & subjects will be clinically assessed for improvement or worsening.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Agreed to participate in this clinical study and signed informed consent, follow-up time greater than 3 months.
3. Comply with the diagnostic criteria of decompensated liver cirrhosis, including liver function damage, portal hypertension clinical manifestations, laboratory and imaging studies.

Exclusion Criteria:

1. Ongoing bacterial infection requiring antibiotic treatment.
2. current or history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening (significant alcohol consumption is defined as more than 20 g/day in females and more than 30 g/day in males, on average).
3. consecutive months within 1 year prior to screening.
4. Treatment with antibiotics or probiotics in the preceding 3 months.
5. Inability to safely perform an GastroIntestinal endoscopy.
6. No history of recent spontaneous bacterial peritonitis or gastrointestinal bleeding.(14 days).
7. Human Immunodeficiency Virus (HIV) infection.
8. Active, serious medical disease with likely life expectancy less than 5 years.
9. Active substance abuse including inhaled or injection drugs in the year prior to screening.
10. pregnancy, planned pregnancy, potential for pregnancy and unwillingness to use effective birth control during the trial, breast feeding.
11. Any other condition which, in the opinion of the investigator, would impede compliance or hinder completion of the study.
12. History of severe (anaphylactic) food allergy.
13. History of gastroparesis or altered gastric motility -
14. Psychiatric disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-03 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events complication rate in all patients in both groups | 3 months
  Adverse events like the general situation, defecate situation and possible clinical events, including: Incidence of new onset upper gastrointestinal bleed in both groups; development of new onset of ascites in both groups.; Number of Spontaneous Bacterial peritonitis cases in both groups. Acute on Chronic Liver failure cases in both groups.

SECONDARY OUTCOMES:
Improvement in liver function test as compared to baseline in both groups. | 3 months
Reduction in systemic inflammatory markers like TNF-α in both groups. | 3 months
Reduction in systemic inflammatory markers like IL-6 in both groups. | 3 months
  Improvement is defined as improvement in Intestinal mucosa structure pre and post treatment.
Reduction in systemic inflammatory markers like serum endotoxins in both groups. | 3 months
Diamine oxidase（DAO） | 3 months
Histological changes in the intestinal biopsy in both groups. | 3 months
Microbiota composition | 3 months
  Deep sequencing of the microbiota at baseline and post-FMT.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-an Li, Ph.D, Study Chair — First Affiliated Hospital of Chengdu Medical College
Locations (1):
- IEC of Chengdu Medical College, Chendu, China

IPD SHARING:
Plan to Share IPD: No